CLINICAL TRIAL: NCT03573245
Title: Tranexamic Acid in Major Orthopedic Surgery: Comparison of 3 Dosage Regimen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CUF Santarém Hospital (Other)
Responsible Party: Principal Investigator, Angela Sa, MD, CUF Santarém Hospital
Other Study IDs: ATX (Tranexamic acid )
Record Dates: First submitted 2018-06-07; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Tranexamic Acid; Knee Osteoarthritis; Ankle Osteoarthritis; Bleeding
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- intra-op single dose: intra-operative single dose of tranexamic acid
  Interventions: Drug: Tranexamic Acid
- intra-op dose and additional dose: intra-operative dose of tranexamic acid and additional dose 3 hours after
  Interventions: Drug: Tranexamic Acid
- intra-op dose and perfusion: intra-operative dose of tranexamic acid followed by a continuous infusion during 6 hours.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid effect on perioperative bleeding in orthopedic surgery

SUMMARY:
Tranexamic acid has been shown to be effective in reducing blood loss and transfusion in orthopedic surgery. It remains unknown the ideal therapeutic regimen. The goal of this study is to compare 3 dosage regimen of tranexamic acid in patients submitted to major orthopedic surgery.

DETAILED DESCRIPTION:
There is ongoing debate, however, around optimal perioperative tranexamic acid dosing, which varies widely.

A large number of studies comparing tranexamic acid to placebo, overall blood loss and transfusion requirements are both reduced by ≈30%. A well designed tranexamic acid trial will provide answers to the best regimen dosage for perioperative tranexamic acid use. It will benefit patients by reducing allogeneic transfusions and their associated risks and costs, thus adding value to the care delivered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 anos
* Total ankle arthroplasty
* Total knee arthroplasty
* Weight >50 kilogram

Exclusion Criteria:

* Allergy and Hypersensitivity to tranexamic acid
* Thromboembolic events history
* Epilepsy
* Acute kidney injury, Glomerular Filtration Rate < 50 ml/min
* Coagulation disorders
* Surgical reintervention
* Blood transfusion refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Patients of a median size private hospital in Portugal
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative bleeding | postoperative day 2
  perioperative blood loss measured in mililiters (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Sa, MD, Principal Investigator — CUF Santarem Hospital

IPD SHARING:
Plan to Share IPD: No